CLINICAL TRIAL: NCT00136942
Title: A Multicenter, 6-Week-Treatment, Open-Label Study Assessing The Percentage Of Hyperlipidemic Patients Achieving Low Density Lipoprotein Cholesterol Target With Atorvastatin
Brief Title: A Swiss Study With Atorvastatin in Hyperlipidemic Patients Measuring LDL-Cholesterol
Acronym: ACTFAST SWISS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2581089
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin

SUMMARY:
The proportion of patients achieving LDL-C target as defined by Swiss cholesterol recommendations (AGLA-recommendations) across starting doses of 10 mg, 20 mg, 40 mg, and 80 mg of atorvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Risk factors and diagnosis of dyslipidemia according to the AGLA-recommendations (see appendix B) at screening
* LDL-C < 6.0 mmol/l
* Triglyceride level < 5.0 mmol/l.

Exclusion Criteria:

* Subjects receiving higher than "usual maintenance" doses of Lipid Lowering Therapy (LLT) at screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370
Dates: Start 2005-04

PRIMARY OUTCOMES:
The proportion of patients achieving LDL-C target as defined by local swiss AGLArecommendations across starting doses of 10 mg, 20 mg, 40 mg, and 80 mg of atorvastatin.

SECONDARY OUTCOMES:
The proportion of patients across different AGLA-categories (primary and secondary prevention) achieving LDL-C target as defined by AGLA-recommendations across starting doses of 10 mg, 20 mg, 40 mg, and 80 mg of atorvastatin.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- Switzerland (20):
  - Pfizer Investigational Site, Binningen, Basel-Landschaft
  - Pfizer Investigational Site, Liestal, Basel-Landschaft
  - Pfizer Investigational Site, Basel, Canton of Basel-City
  - Pfizer Investigational Site, Langenthal, Canton of Bern
  - Pfizer Investigational Site, Thun, Canton of Bern
  - Pfizer Investigational Site, Düdingen, Canton of Fribourg
  - Pfizer Investigational Site, Geneva, Canton of Geneva
  - Pfizer Investigational Site, Onex, Canton of Geneva
  - Pfizer Investigational Site, Pfaeffikon, Canton of Schwyz
  - Pfizer Investigational Site, Siebnen, Canton of Schwyz
  - Pfizer Investigational Site, Écublens, Canton of Vaud
  - Pfizer Investigational Site, Lausanne, Canton of Vaud
  - Pfizer Investigational Site, Prilly, Canton of Vaud
  - Pfizer Investigational Site, Unterägeri, Canton of Zug
  - Pfizer Investigational Site, Zug, Canton of Zug
  - Pfizer Investigational Site, Zurich, Canton of Zurich
  - Pfizer Investigational Site, Lugano, Canton Ticino
  - Pfizer Investigational Site, Malvaglia, Canton Ticino
  - Pfizer Investigational Site, Melide, Canton Ticino
  - Pfizer Investigational Site, Vezia, Canton Ticino

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581089&StudyName=ACTFAST+Swiss%3A+a+Swiss+Study+with+Atorvastatin+in+Hyperlipidemic+Patients+measuring+LDL%2DCholesterol